CLINICAL TRIAL: NCT03355170
Title: Cardiac Safety Evaluation of Lansoprazole/Domperidone 30/30 mg Sustained Release Capsule Formulation
Brief Title: Cardiac Safety of Lansoprazole and Domperidon Combination
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The sponsor decided to continue with a different design and a different protocol.
Sponsor: Neutec Ar-Ge San ve Tic A.Ş (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: NEU-05.16
Record Dates: First submitted 2017-11-20; First posted 2017-11-28 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: GERD; Cardiac Event; Safety Issues
MeSH Terms: conditions — Gastroesophageal Reflux; Cardiovascular Diseases | interventions — Lansoprazole; Domperidone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lansoprazole/Domperidone (Experimental): Patient will be administered lansoprazole/domperidone 30/30 mg capsules (brand name: Duolans) half an hour before breakfast for eight weeks according to randomisation scheme.
  Interventions: Combination Product: Lansoprazole/Domperidone
- Lansoprazole (Active Comparator): Patient will be administered lansoprazole 30 mg capsules (brand name: Lasotab) half an hour before breakfast for eight weeks according to randomisation scheme.
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Combination Product: Lansoprazole/Domperidone — Experimental
  Other Names: Duolans
  Arms: Lansoprazole/Domperidone
Drug: Lansoprazole — Active comparator
  Other Names: Lasotab
  Arms: Lansoprazole

SUMMARY:
The aim of current study is to compare safety and efficacy of lansoprazole/domperidone 30/30 mg sustained release capsules (brand name: Duolans) and lansoprazole 30 mg micropellet capsules (brand name: Lasotab) in GERD patients in terms of cardiac safety.

ELIGIBILITY:
Inclusion Criteria:

* GERD patients with BMI 18-33 kg/m2
* Patients with esophagitis class A-B according to Los Angeles classification

Exclusion Criteria:

* Patients whose long QT syndrome risk score > 3.
* Patients with family history of short or long QT syndrome.
* Patients with Barrett's stricture, gastric outlet obstruction, malignancy, gastrointestinal system bleeding or any other upper gastrointestinal system pathology.
* Patients whose Hiatus hernia is > 3 cm.
* Patients with uncontrolled or insulin dependent diabetes mellitus, symptomatic gallbladder stone, active or unhealed stomach or duodenum ulcer, Zollinger-Ellison syndrome, primary esophagus motility disorder, pancreatitis, inflammatory bowel disease, severe lung disease, chronic liver disease, uncontrolled kidney impairment, cancer (except skin cancer except melanoma), cerebrovascular disease, epilepsy.
* Patients with history of heart failure, ventricular tachycardia, ventricular fibrillation, cardiac arrest, Torsades de pointes, bradycardia, sinus node dysfunction, heart attack, long QTc (>460 ms).
* Patients taken PPIs or H2-blockers within 7 days and prokinetic drugs within 3 days before entering the study.
* Patients with major psychiatric disease.
* Alcoholism and drug use.
* Patients with pathologic laboratory tests; hemogram, sedimentation, CRP, thyroid functions tests, liver enzymes.
* Malabsorption.
* Immunosuppressive patients.
* Patients taken cortisone.
* Patients taken other drugs that prolong QT interval.
* Patients taken drugs that need gastric acid for optimal absorption; ketoconazole, iron salts, digoxin, ampicillin esters, anticoagulants, antineoplastic agents, prostaglandin analogues, sucralfate, atazanavir, theophylline, tacrolimus, fluvoxamine, rifampisin, nefazodone and aprepitant.
* Patients taken drugs carried with P-glycoprotein, indicated for heart diseases, AIDS/HIV or infection treatment.
* Pregnancy or breast-feeding.
* Patients taken drugs that may affect gastrointestinal system motility or acid release.
* History of abdominal surgery (hysterectomy, abdominal hernia repair, caesarean cases may be included; cholecystectomy have to be excluded).
* Patients with hypocalcemia and hypercalcemia
* Patients taken NSAII drugs (paracetamol may be used up to 2 gr/day).
* Patients taken antidepressants.
* Hypersensitivity to study drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2018-12-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Change in QT and corrected QT (QTc) interval compared to baseline | 8 weeks

SECONDARY OUTCOMES:
Change in upper gastrointestinal symptom severity index compared to baseline. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Serhat Bor, Prof Dr, Study Chair — Ege University Medical Faculty Gastroenterology Dep.
Locations (16):
- Turkey (Türkiye) (16):
  - Başkent University Hospital Gastroenterology Dep., Adana
  - Çukurova University Medical Faculty Cardiology Dep., Adana
  - Ankara University Medical Faculty Gastroenterology Dep., Ankara
  - Dışkapı Research and Training Hospital Gastroenterology Dep., Ankara
  - Yüksek İhtisas Research and Training Hospital Gastroenterology Dep., Ankara
  - Antalya Research and Training Hospital Gastroenterology Dep., Antalya
  - Balıkesir University Medical Faculty Gastroenterology Dep., Balıkesir
  - Gaziantep Şahinbey Research and Training Hospital Gastroenterology Dep., Gaziantep
  - Dr. Sadi Konuk Research and Training Hospital Gastroenterology Dep., Istanbul
  - Ümraniye Research and Training Hospital Gastroenterology Dep., Istanbul
  - Ege University Medical Faculty Gastroenterology Dep., Izmir
  - Tepecik Research and Training Hospital Gastroenterology Dep., Izmir
  - Celal Bayar University Medical Faculty Gastroenterology Dep., Manisa
  - Sıtkı Koçman University Medical Faculty Gastroenterology Dep., Muğla
  - Recep Tayyip Erdoğan University Medical Faculty Gastroenterology Dep., Rize
  - Cumhuriyet University Medical Faculty Gastroenterology Dep., Sivas

IPD SHARING:
Plan to Share IPD: No